CLINICAL TRIAL: NCT06278168
Title: Raising Awareness of Autism Spectrum Disorder in Children: Promoting Understanding and Support
Brief Title: Awareness Training in Children With Autism Spectrum Disorder.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2024-002
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; children; ASD; awareness
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental awareness group (Experimental): Twenty children in the experimental group will undergo individual training in which they will watch relaxation videos with the Oculus device. The group sessions will be the same for both groups.
  Interventions: Other: Awareness training with using Oculus.
- Traditional awareness group (Other): Twenty children in the control group will undergo individual training without using Oculus device. The group sessions will be the same for both groups.
  Interventions: Other: Awareness training without using Oculus

INTERVENTIONS:
Other: Awareness training with using Oculus. — The protocol consists of 2 phases:one conducted in groups,one individually. In the first session, through interactive activities such as passing a wool ball while sharing passions and interests, and filling out personal cards, participants get to know each other and develop an atmosphere of mutual acceptance.
  In the second session,participants explore neurodiversity through viewing videos, guided discussions and creating symbols representative of the group concept. Optical illusions are explored to understand differences in individual perception.In addition, issues of hypersensitivity and hyposensitivity are addressed,encouraging participants to reflect on their special interests and ways of presenting themselves. The second phase consists of 12 individual meetings to promote emotional well-being and self-awareness. During the meetings, the Oculus device will be used in which relaxation videos will be shown. In addition, heart rate will be detected with sensors placed in the chest.
  Arms: Experimental awareness group
Other: Awareness training without using Oculus — The control group will carry out the same steps as the experimental group, heart rate will be taken through the use of sensors but in this case the Oculus device will not be used to watch relaxation videos.
  Arms: Traditional awareness group

SUMMARY:
The proposed protocol aims to facilitate awareness and understanding of autism spectrum disorder among children aged 8 to 14 with an IQ between 85 and 115. Conducted once a week for 60 minutes, the protocol encompasses two initial group sessions followed by 5 group meetings, introducing activities to foster self-awareness, cognitive understanding, and an inclusive environment. Subsequently, the protocol advances to 12 individual sessions focused on emotional well-being and self-awareness, integrating Oculus technology and chest sensors for heart rate monitoring. Initiating the intervention, individual family meetings are scheduled to outline intervention goals and phases. The initial group sessions focus on social bonding, cognitive understanding, and creating an accepting atmosphere among participants. Utilizing activities addressing neurodiversity awareness and technological tools like tablets, the sessions encourage discussions on individual differences and sensitivities. The subsequent individual sessions are structured to explore personal values, identify inner critical voices, and develop emotional awareness through exercises exploring emotions and physical sensations. Progressively, the intervention introduces mindfulness, guiding participants to acknowledge emotions as normal and encouraging alignment of daily actions with personal values. Following this, sessions center on building observational skills, recognizing past behaviors, and fostering strengths tied to values. Participants are encouraged to distinguish between their critical "consultant" and the value-driven "explorer," fostering personal growth and reflection. The protocol's later stages delve into identifying personal strengths linked to core values and exploring value-driven goals. Visual exercises, metaphors, and flexible self-views are emphasized, promoting adaptability and self-evolution. The protocol concludes by advocating a flexible self-view, embracing change, and connecting oneself to ever-evolving metaphors like "a cup with changing contents" or "the ever-changing sky." These sessions culminate with visual relaxation facilitated through Oculus technology while simultaneously monitoring participants' heart rates using chest sensors. This comprehensive approach integrates technological tools with emotional and cognitive exercises, providing a multifaceted framework to enhance self-awareness and promote acceptance within the context of neurodiversity.

ELIGIBILITY:
Inclusion Criteria:

* 85<IQ<115

Exclusion Criteria:

* presence of other medical disorders

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-05-08 (Estimated)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children Fourth edition (WISC-IV) | The test needs approximately 65-80 minutes to complete.
  Wechsler Intelligence Scale for Children Fourth edition (WISC-IV) is a clinical tool for assessing the cognitive abilities of children and young people between the ages of 6 years and 16 years and 11 months.
  The WISC-IV scales are as follows: index of verbal comprehension (ICV), range weighted scores (min 46 - max154); index visuoperceptual reasoning (IRP), range weighted scores (min 41- max 159); index working memory (IML) range weighted scores (min 46 - max 154); processing speed index (IVE) range weighted scores (min 47 - max 153); intelligence quotient IQ (min 40 - max
  160). For each sub-scale higher score corresponds to better performance.
Multidimensional Anxiety Scale for Children-Second Edition (MASC 2) | The test needs approximately 15 minutes
  MASC 2 is an assessment tool for anxiety-related symptoms consisting of a self-report questionnaire and rating scales for parents. it consists of 50 items.
Screen for Child Anxiety Related Disorders (SCARED) | The estimated time for administration of this sub-test is about 10-15 minutes.
  The SCARED - Screen for child Anxiety Related Emotional Disorders questionnaire is considered one of the best tools for measuring childhood anxiety. The SCARED is a child and parent self-report instrument used to screen for childhood anxiety disorders including general anxiety disorder, separation anxiety disorder, panic disorder, and social phobia. Also, evaluate symptoms related to school phobias.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Bruin EI, Blom R, Smit FM, van Steensel FJ, Bogels SM. MYmind: Mindfulness training for Youngsters with autism spectrum disorders and their parents. Autism. 2015 Nov;19(8):906-14. doi: 10.1177/1362361314553279. Epub 2014 Oct 27. PMID 25348866
- [Background] Louise L.Hayes, Joseph Ciarrochi (2015). Adolescenti in crescita. L'ACT per aiutare i giovani a gestire le emozioni, raggiungere obiettivi, costruire relazioni sociali. Franco Angeli